CLINICAL TRIAL: NCT03822832
Title: Phase IIa, Multicentre, Randomized, Double-blind, Placebo-controlled, Study to Evaluate the Safety, Tolerability and Efficacy of Treatment With BI 655130 in Adult Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study in Patients With Atopic Eczema to Test How Effective BI 655130 is and How Well it is Tolerated
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1368-0032
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Results first posted 2022-12-01 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — spesolimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Spesolimab (Experimental): i.v.
  Interventions: Drug: BI 655130
- Placebo (Placebo Comparator): i.v.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 655130 — Solution for infusion
  Other Names: Spesolimab
  Arms: Spesolimab
Drug: Placebo — Solution for infusion
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to investigate the safety, tolerability and efficacy of BI 655130 in patients with Atopic Dermatitis (AD) following repeated intravenous administrations compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent in accordance with Good Clinical Practice (GCP) and local legislation prior to the start of any screening procedures
* Male or female patients, 18 to 75 years of age at screening
* Diagnosis of atopic dermatitis for at least 1 year
* Moderate to severe atopic dermatitis defined as:

  * At least 10% Body Surface Area (BSA) of atopic dermatitis involvement at screening and baseline
  * Eczema Area and Severity Index (EASI) of at least 12 at screening and at least 16 at baseline
  * Investigator Global Assessment (IGA) of at least 3 at screening and baseline
* Documented history of inadequate response to topical corticosteroid as judged by the investigator
* Willing to use a standard emollient for the duration of the study
* Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.

Exclusion Criteria:

* Use of topical corticosteroids or other agents for atopic dermatitis within 7 days prior to first dose of trial treatment.
* Use of systemic corticosteroids or other agents for atopic dermatitis within 4 weeks prior to first dose of trial treatment.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial. Women who stop nursing before the study drug administration do not need to be excluded from participating; they should refrain from breastfeeding up to 16 weeks after the last study drug administration
* Patient with a transplanted organ (with exception of a corneal transplant > 12 weeks prior to screening) or who have ever received stem cell therapy (e.g., Prochymal).
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to the screening visit, except appropriately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix.
* Use of any restricted medication or any drug considered likely to interfere with the safe conduct of the study, as assessed by the investigator.
* History of allergy/hypersensitivity to the systemically administered trial medication agent or its excipients.
* Active systemic infections (Fungal and bacterial disease) during the last 2 weeks prior to first drug administration, per investigator assessment.
* Relevant chronic or acute infections (exception: common cold) including human immunodeficiency virus (HIV) or viral hepatitis. A patient can be re-screened if the patient was treated and is cured from the acute infection.
* Active or Latent Tuberculosis (TB):

  * Patients with active tuberculosis are excluded.
  * Patients with a positive QuantiFERON TB test during screening are excluded, unless:

    * Patient had previous diagnosis of active or latent TB and has completed appropriate treatment per local practice/guidelines within the last 3 years and at least 6 months before first administration of trial medication under this protocol (patients may be re-screened once to meet this criterion)
    * Patients with suspected false positive or indeterminate QuantiFERON TB result may be re-tested once
    * If the QuantiFERON TB test result is not available or provides indeterminate results after repeat testing: A tuberculin skin test reaction ≥10mm (≥5mm if receiving ≥15mg/d prednisone or its equivalent) is considered positive.
* Currently enrolled in another investigational device or drug trial, or less than 30 days or 5 half lives, whichever is longer since ending another investigational device or drug trial(s), or receiving other investigational treatment(s).
* Evidence of a current or previous disease, medical condition (including chronic alcohol or drug abuse or any condition) other than AD, surgical procedure, psychiatric or social problems, medical examination finding (including vital signs and ECG), or laboratory value at the screening outside the reference range that in the opinion of the investigator is clinically significant and would make the study participant unreliable to adhere to the protocol, comply with all study visits/procedures or to complete the trial, compromise the safety of the patient or compromise the quality of the data.
* Major surgery (major according to the investigator) performed within 12 weeks prior to first study drug adminstration or planned during the study (e.g. hip replacement, aneurysm removal, stomach ligation).
* Severe, progressive, or uncontrolled hepatic disease, defined as >3-fold Upper Limit of Normal (ULN) elevation in AST or ALT or alkaline phosphatase, or >2-fold ULN elevation in total bilirubin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-07-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (10):
  - Center for Dermatology and Plastic Surgery, Scottsdale, Arizona
  - Clinical Physiology Associates, Fort Myers, Florida
  - Finlay Medical Research Corp, Miami, Florida
  - University of South Florida, Tampa, Florida
  - ForCare Clinical Research, Inc., Tampa, Florida
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Dermatology Treatment and Research Center, PA, Dallas, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
- Canada (3):
  - University of Alberta Hospital (University of Alberta), Edmonton, Alberta
  - NewLab Clinical Research Inc., St. John's, Newfoundland and Labrador
  - Innovaderm Research Inc., Montreal, Quebec
- Japan (10):
  - Aichi Medical University Hospital, Aichi, Nagakute
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Kurume University Hospital, Fukuoka, Kurume
  - Hosui General Medical Clinic, Hokkaido, Sapporo
  - Tennocho Ekimae Dermatology and Allergology, Kanagawa, Yokohama
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Osaka City University Hospital, Osaka, Osaka
  - Tokyo Medical University Hachioji Medical Center, Tokyo, Hachioji
  - Showa University Hospital, Tokyo, Shinagawa-ku

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Lebwohl MG, Thoma C, Haeufel T. Spesolimab use in generalised pustular psoriasis flares - Authors' reply. Lancet. 2024 Aug 31;404(10455):847-848. doi: 10.1016/S0140-6736(24)01557-5. No abstract available. PMID 39216969
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase IIa multicentre, randomized, double-blind, placebocontrolled, study to evaluate the safety, tolerability and efficacy of treatment with BI 655130 in adult patients with moderate to severe atopic dermatitis.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo Intravenous Every 4 Weeks: Placebo intravenous (i.v.) infusion once every 4 weeks (q4w) during the double blind period from week 0 to 16 (4 treatments in total). At week 16 patients were assessed based on their Eczema Area and Severity Index (EASI) score, patients with EASI≥75 were classified as responders and patients with EASI<75 were classified as non-responders. Responders received no further treatment, non-responders were offered an open label treatment with 600 mg Spesolimab (BI 655130) i.v. infusion once every 4 weeks from week 16 to 28 (4 treatments in total, last dose at week 28). End of study was at week 44.
- Spesolimab 600 mg Intravenous Every 4 Weeks: 600 milligram (mg) Spesolimab (BI 655130) intravenous (i.v.) infusion once every 4 weeks (q4w) during the double blind period from week 0 to 16 (4 treatments in total). At week 16 patients were assessed based on their Eczema Area and Severity Index (EASI) score, patients with EASI≥75 were classified as responders and patients with EASI<75 were classified as non-responders. Responders received no further treatment, non-responders were offered an open label treatment with 600 mg Spesolimab (BI 655130) i.v. infusion once every 4 weeks from week 16 to 28 (4 treatments in total, last dose at week 28). End of study was at week 44.
Period: Period 1 - Double Blind Period
Arm/Group | Placebo Intravenous Every 4 Weeks | Spesolimab 600 mg Intravenous Every 4 Weeks
Started | 18 | 33
Completed | 8 | 22
Not Completed | 10 | 11
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Lack of Efficacy | 2 | 1
Not completed — Adverse Event | 3 | 5
Period: Re-allocation
Arm/Group | Placebo Intravenous Every 4 Weeks | Spesolimab 600 mg Intravenous Every 4 Weeks
Started | 8 | 22
Completed (Patient re-allocated to open label Spesolimab treatment) | 6 (Patient re-allocated to open label Spesolimab treatment) | 16 (Patient re-allocated to open label Spesolimab treatment)
Not Completed | 2 | 6
Not completed — Not re-allocated to open label period | 2 | 6
Period: Period 2 - Open Label Period
Arm/Group | Placebo Intravenous Every 4 Weeks | Spesolimab 600 mg Intravenous Every 4 Weeks
Started | 6 (Patient re-allocated to open label Spesolimab treatment) | 16 (Patient re-allocated to open label Spesolimab treatment)
Completed | 5 | 13
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 0 | 3

BASELINE CHARACTERISTICS:
Population: Randomized set (RS): this patient set includes all patients who were randomized into the trial. It will be used for display of patient disposition, baseline and demographic characteristics, and patients with IPDs (Important Protocol Deviations).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Intravenous Every 4 Weeks | Spesolimab 600 mg Intravenous Every 4 Weeks | Total
Number analyzed (Participants) | 18 | 33 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (12.4) | 43.2 (15.9) | 39.4 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 7 | 18 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 15 | 27 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 10 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 7 | 17 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: Score on a scale] — Eczema Area and Severity Index (EASI) Score assesses the extent of disease at four body sites and measures four clinical signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification, each on a scale of zero to three. The EASI score confers a maximum of 72 and evaluates two dimensions of Atopic Dermatitis (AD): disease extent and clinical signs. The suggested severity strata for the EASI are as follows: 0 = clear; 0.1-1.0 = almost clear; 1.1-7.0 = mild; 7.1-21.0 = moderate; 21.1-50.0 = severe; 50.1-72.0 = very severe.
  Score on a scale | 26.43 (8.60) | 26.53 (10.07) | 26.50 (9.49)
SCORing of Atopic Dermatitis (SCORAD) [Mean (Standard Deviation); unit: Score on a scale] — SCORing of Atopic Dermatitis (SCORAD). Extent (A): rule of 9 was used to calculate body surface area affected by AD. The score for each body region was added to A (0-100). Intensity (B): intensity of each sign was assessed from none=0 to severe=3. Scores summed to B (0-18). Subjective symptoms (C): pruritus and sleep loss, each of these 2 were scored using visual analogue scale from 0 to 10, higher scores=worse. Scores for itch and sleeplessness were added to give 'C' (0-20). The SCORAD for an individual was calculated: A/5 + 7*B/2 + C; range from 0 to 103; higher values of SCORAD=worse.
  Score on a scale | 62.82 (14.13) | 60.09 (10.36) | 61.06 (11.76)
Investigator's Global Assessment (IGA) score [Mean (Standard Deviation); unit: Score on a scale] — Investigator's Global Assessment (IGA) score allows investigators to assess the overall disease severity at one given time point. It is a 5-point scale with: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe. The overall IGA score includes the assessment of erythema, induration/papulation, lichenification, and oozing/crusting. For the first three sections the following scale will be used: "None", "Barely Perceptible" ("Minimal" for lichenification), "Slight but Definite", "Clearly Perceptible" or "Marked". For oozing/crusting the available answers are "None" or "Present."
  Score on a scale | 3.4 (0.5) | 3.2 (0.4) | 3.3 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in the Eczema Area and Severity Index (EASI) Score at Week 16
Description: Percentage change from baseline in the Eczema Area and Severity Index (EASI) Score at Week 16. The EASI score assesses the extent of disease at four body sites and measures four clinical signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification, each on a scale of zero to three. The EASI score confers a maximum of 72 and evaluates two dimensions of Atopic Dermatitis (AD): disease extent and clinical signs. The suggested severity strata for the EASI are as follows: 0 = clear; 0.1-1.0 = almost clear; 1.1-7.0 = mild; 7.1-21.0 = moderate; 21.1-50.0 = severe; 50.1-72.0 = very severe.
  Restricted maximum likelihood(REML)-based Mixed Model Repeated Measures (MMRM) including fixed, categorical effects of treatment, visit, and Asian/Non-Asian (yes/no) as well as the treatment-by-visit interaction, and continuous, fixed covariates of baseline endpoint and baseline-by-visit interaction. Unstructured covariance matrix was used.
Time Frame: Baseline (day 1) and Week 16 (day 113 ±3 days), up to 116 days.
Population: Full Analysis Set (FAS): All participants who were randomised, received at least one dose during the trial, and had a baseline measurement for the primary endpoint.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo Intravenous Every 4 Weeks | Spesolimab 600 mg Intravenous Every 4 Weeks
Number analyzed (Participants) | 12 | 28
Percent change | -12.3 (14.3) | -37.9 (9.8)
Statistical Analysis 1: Comparison: Placebo Intravenous Every 4 Weeks vs Spesolimab 600 mg Intravenous Every 4 Weeks; Test type: Other; p = 0.1492, Mixed Models Analysis; See endpoint description for model description; Mean Difference (Final Values) = -25.6, 90% CI 2-sided [-54.9 to 3.7], Standard Error of Mean 17.4 — Difference calculated as Spesolimab - Placebo

2. Secondary Outcome: Number of Patients With Drug Related Adverse Events (AEs)
Description: Number of patients with drug related Adverse Events (AEs) reported separately in both for the double blind period as well as the re-allocation treatment period.
  Double blind period: Baseline (week 1) to the last study drug administration date (week 12) + Residual effects period (REP, 16 weeks). For patients who initiated the re-allocation treatment period the REP was shortened to the date of first re-allocation treatment period treatment administration. Up to a total time frame of 28 weeks.
  Re-allocation treatment period: Week 1 of re-allocation treatment period to the last study drug administration date (week 12 of re-allocation treatment period) + REP (16 weeks), or end-of-study date, whichever occurred earlier. Up to a total time frame of 28 weeks.
Time Frame: Up to 28 weeks, see endpoint description for more details.
Population: Double blind period: Safety Analysis Set (SAF): patients who were randomised, and received at least one dose during the trial.
  Re-allocation treatment period: This patient set includes all randomized patients who received at least one dose of study drug and received study medication after re-allocation visit (i.e., after Week 16 visit).
Measure: Number; unit: Participants
Arm/Group | Placebo Intravenous Every 4 Weeks | Spesolimab 600 mg Intravenous Every 4 Weeks
Number analyzed (Participants) | 18 | 33
Participants
  Double blind treatment period | 6 | 4
  Re-allocation treatment period: number analyzed (Participants) | 6 | 16
  Re-allocation treatment period | 0 | 2

3. Secondary Outcome: Absolute Change From Baseline in Eczema Area and Severity Index (EASI) at Week 4
Description: Absolute change from baseline in the Eczema Area and Severity Index (EASI) Score at Week 4. The EASI score assesses the extent of disease at four body sites and measures four clinical signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification, each on a scale of zero to three. The EASI score confers a maximum of 72 and evaluates two dimensions of Atopic Dermatitis (AD): disease extent and clinical signs. The suggested severity strata for the EASI are as follows: 0 = clear; 0.1-1.0 = almost clear; 1.1-7.0 = mild; 7.1-21.0 = moderate; 21.1-50.0 = severe; 50.1-72.0 = very severe.
  Restricted maximum likelihood(REML)-based Mixed Model Repeated Measures (MMRM) including fixed, categorical effects of treatment, visit, and Asian/Non-Asian (yes/no) as well as the treatment-by-visit interaction, and continuous, fixed covariates of baseline endpoint and baseline-by-visit interaction. Unstructured covariance matrix was used.
Time Frame: Baseline (day 1) and Week 4 (day 29 ±3 days), up to 32 days.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Change in score on a scale
Arm/Group | Placebo Intravenous Every 4 Weeks | Spesolimab 600 mg Intravenous Every 4 Weeks
Number analyzed (Participants) | 16 | 29
Change in score on a scale | -7.0 (3.0) | -6.3 (2.2)
Statistical Analysis 1: Comparison: Placebo Intravenous Every 4 Weeks vs Spesolimab 600 mg Intravenous Every 4 Weeks; Test type: Other; p = 0.8613, Mixed Models Analysis; See endpoint description for model description; Mean Difference (Final Values) = 0.7, 90% CI 2-sided [-5.7 to 7.0], Standard Error of Mean 3.8 — Difference calculated as Spesolimab - Placebo

4. Secondary Outcome: Percentage Change From Baseline in Eczema Area and Severity Index (EASI) at Week 4
Description: Percentage change from baseline in the Eczema Area and Severity Index (EASI) Score at Week 4. The EASI score assesses the extent of disease at four body sites and measures four clinical signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification, each on a scale of zero to three. The EASI score confers a maximum of 72 and evaluates two dimensions of Atopic Dermatitis (AD): disease extent and clinical signs. The suggested severity strata for the EASI are as follows: 0 = clear; 0.1-1.0 = almost clear; 1.1-7.0 = mild; 7.1-21.0 = moderate; 21.1-50.0 = severe; 50.1-72.0 = very severe.
  Restricted maximum likelihood(REML)-based Mixed Model Repeated Measures (MMRM) including fixed, categorical effects of treatment, visit, and Asian/Non-Asian (yes/no) as well as the treatment-by-visit interaction, and continuous, fixed covariates of baseline endpoint and baseline-by-visit interaction. Unstructured covariance matrix was used.
Time Frame: Baseline (day 1) and Week 4 (day 29 ±3 days), up to 32 days.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo Intravenous Every 4 Weeks | Spesolimab 600 mg Intravenous Every 4 Weeks
Number analyzed (Participants) | 16 | 29
Percent change | -21.6 (11.3) | -23.8 (8.3)
Statistical Analysis 1: Comparison: Placebo Intravenous Every 4 Weeks vs Spesolimab 600 mg Intravenous Every 4 Weeks; Test type: Other; p = 0.8754, Mixed Models Analysis; See endpoint description for model description; Mean Difference (Final Values) = -2.2, 90% CI 2-sided [-25.8 to 21.4], Standard Error of Mean 14.0 — Difference calculated as Spesolimab - Placebo

5. Secondary Outcome: Proportion of Patients With a 50% Improvement From Baseline in Eczema Area and Severity Index (EASI)(EASI50) at Week 4 and 16
Description: Proportion of patients with a 50% improvement from baseline in Eczema Area and Severity Index (EASI)(EASI50) at Week 4 and 16. The EASI score assesses the extent of disease at four body sites and measures four clinical signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification, each on a scale of zero to three. The EASI score confers a maximum of 72 and evaluates two dimensions of Atopic Dermatitis (AD): disease extent and clinical signs. The suggested severity strata for the EASI are as follows: 0 = clear; 0.1-1.0 = almost clear; 1.1-7.0 = mild; 7.1-21.0 = moderate; 21.1-50.0 = severe; 50.1-72.0 = very severe.
Time Frame: Baseline (day 1) and Week 16 (day 113 ±3 days), up to 116 days.
Population: as for outcome 1
Measure: Number; unit: Proportion of patients
Arm/Group | Placebo Intravenous Every 4 Weeks | Spesolimab 600 mg Intravenous Every 4 Weeks
Number analyzed (Participants) | 18 | 33
Proportion of patients
  Week 4 | 0.333 | 0.303
  Week 16 | 0.056 | 0.303
Statistical Analysis 1: Comparison: Placebo Intravenous Every 4 Weeks vs Spesolimab 600 mg Intravenous Every 4 Weeks; Risk difference at week 4; Test type: Other; CIs are calculated using the method of Wilson and Newcombe; Risk Difference (RD) = -0.030, 90% CI 2-sided [-0.254 to 0.176] — Difference calculated as Spesolimab - Placebo
Statistical Analysis 2: Comparison: Placebo Intravenous Every 4 Weeks vs Spesolimab 600 mg Intravenous Every 4 Weeks; Risk difference at week 16; Test type: Other; CIs are calculated using the method of Wilson and Newcombe; Risk Difference (RD) = 0.247, 90% CI 2-sided [0.053 to 0.396] — Difference calculated as Spesolimab - Placebo

6. Secondary Outcome: Proportion of Patients With a 75% Improvement From Baseline in Eczema Area and Severity Index (EASI)(EASI75) at Week 4 and 16
Description: Proportion of patients with a 75% improvement from baseline in Eczema Area and Severity Index (EASI)(EASI75) at Week 4 and 16. The EASI score assesses the extent of disease at four body sites and measures four clinical signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification, each on a scale of zero to three. The EASI score confers a maximum of 72 and evaluates two dimensions of Atopic Dermatitis (AD): disease extent and clinical signs. The suggested severity strata for the EASI are as follows: 0 = clear; 0.1-1.0 = almost clear; 1.1-7.0 = mild; 7.1-21.0 = moderate; 21.1-50.0 = severe; 50.1-72.0 = very severe.
Time Frame: Baseline (day 1) and Week 16 (day 113 ±3 days), up to 116 days.
Population: as for outcome 1
Measure: Number; unit: Proportion of patients
Arm/Group | Placebo Intravenous Every 4 Weeks | Spesolimab 600 mg Intravenous Every 4 Weeks
Number analyzed (Participants) | 18 | 33
Proportion of patients
  Week 4 | 0.111 | 0.091
  Week 16 | 0.056 | 0.152
Statistical Analysis 1: Comparison: Placebo Intravenous Every 4 Weeks vs Spesolimab 600 mg Intravenous Every 4 Weeks; Risk difference at week 4; Test type: Other; CIs are calculated using the method of Wilson and Newcombe; Risk Difference (RD) = -0.020, 90% CI 2-sided [-0.204 to 0.117] — Difference calculated as Spesolimab - Placebo
Statistical Analysis 2: Comparison: Placebo Intravenous Every 4 Weeks vs Spesolimab 600 mg Intravenous Every 4 Weeks; Risk difference at week 16; Test type: Other; CIs are calculated using the method of Wilson and Newcombe; Risk Difference (RD) = 0.096, 90% CI 2-sided [-0.080 to 0.232] — Difference calculated as Spesolimab - Pl

7. Secondary Outcome: Change From Baseline in SCORing of Atopic Dermatitis (SCORAD) at Week 4
Description: SCORing of Atopic Dermatitis (SCORAD). Extent (A): rule of 9 was used to calculate body surface area affected by AD. The score for each body region was added to determine A (0-100). Severity (B): severity of each sign (erythema; edema; oozing; excoriation; skin thickening; dryness) was assessed from none=0to severe=3. Severity scores summed to B (0-18). Subjective symptoms (C): pruritus and sleep, each of these 2 were scored by participant/caregiver using visual analogue scale from 0 to 10, higher scores=worse symptoms. Scores for itch and sleeplessness were added to give 'C' (0-20). The SCORAD for an individual was calculated: A/5 + 7*B/2 + C; range from 0 to 103; higher values of SCORAD=worse outcome.
  REML-based MMRM including fixed, categorical effects of treatment, visit, and Asian/Non-Asian as well as the treatment-by-visit interaction, and continuous, fixed covariates of baseline endpoint and baseline-by-visit interaction. Unstructured covariance matrix was used.
Time Frame: Baseline (day 1) and Week 4 (day 29 ±3 days), up to 32 days.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Change in score on a scale
Arm/Group | Placebo Intravenous Every 4 Weeks | Spesolimab 600 mg Intravenous Every 4 Weeks
Number analyzed (Participants) | 16 | 29
Change in score on a scale | -13.3 (7.0) | -13.2 (5.2)
Statistical Analysis 1: Comparison: Placebo Intravenous Every 4 Weeks vs Spesolimab 600 mg Intravenous Every 4 Weeks; Test type: Other; p = 0.9900, Mixed Models Analysis; See endpoint description for model description; Mean Difference (Final Values) = 0.1, 90% CI 2-sided [-14.6 to 14.8], Standard Error of Mean 8.7 — Difference calculated as Spesolimab - Placebo

8. Secondary Outcome: Change From Baseline in SCORing of Atopic Dermatitis (SCORAD) at Week 16
Description: as for outcome 7
Time Frame: Baseline (day 1) and Week 16 (day 113 ±3 days), up to 116 days.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Change in score on a scale
Arm/Group | Placebo Intravenous Every 4 Weeks | Spesolimab 600 mg Intravenous Every 4 Weeks
Number analyzed (Participants) | 12 | 28
Change in score on a scale | -10.7 (10.0) | -25.5 (6.8)
Statistical Analysis 1: Comparison: Placebo Intravenous Every 4 Weeks vs Spesolimab 600 mg Intravenous Every 4 Weeks; Test type: Other; p = 0.2266, Mixed Models Analysis; See endpoint description for model description; Mean Difference (Final Values) = -14.9, 90% CI 2-sided [-35.2 to 5.5], Standard Error of Mean 12.1 — Difference calculated as Spesolimab - Placebo

9. Secondary Outcome: Number of Patients Achieving at Least a 2-grade Reduction From Baseline to Clear (0) or Almost Clear (1) in Investigator's Global Assessment (IGA) at Week 4 and 16
Description: Number of patients achieving at least a 2-grade reduction from baseline to clear (0) or almost clear (1) in Investigator's Global Assessment (IGA) at Week 4 and 16. IGA score allows investigators to assess the overall disease severity at one given time point. It is a 5-point scale with: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe. The overall IGA score includes the assessment of erythema, induration/papulation, lichenification, and oozing/crusting. For the first three sections the following scale will be used: "None", "Barely Perceptible" ("Minimal" for lichenification), "Slight but Definite", "Clearly Perceptible" or "Marked". For oozing/crusting the available answers are "None" or "Present."
Time Frame: Baseline (day 1) and Week 16 (day 113 ±3 days), up to 116 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Intravenous Every 4 Weeks | Spesolimab 600 mg Intravenous Every 4 Weeks
Number analyzed (Participants) | 18 | 33
Participants
  Week 4 | 1 | 2
  Week 16 | 0 | 3
Statistical Analysis 1: Comparison: Placebo Intravenous Every 4 Weeks vs Spesolimab 600 mg Intravenous Every 4 Weeks; Risk difference at week 4; Test type: Other; CIs are calculated using the method of Wilson and Newcombe; Risk Difference (RD) = 0.005, 90% CI 2-sided [-0.159 to 0.120] — Difference calculated as Spesolimab - Placebo
Statistical Analysis 2: Comparison: Placebo Intravenous Every 4 Weeks vs Spesolimab 600 mg Intravenous Every 4 Weeks; Risk difference at week 16; Test type: Other; CIs are calculated using the method of Wilson and Newcombe; Risk Difference (RD) = 0.091, 90% CI 2-sided [-0.050 to 0.207] — Difference calculated as Spesolimab - Placebo

ADVERSE EVENTS:
Time Frame: Double blind period: Baseline to the last study drug administration date + REP (16 weeks). For patients who initiated the open label treatment the REP was shortened to the date of first open label treatment administration. Up to a total time frame of 28 weeks. Open label period: Week 16 to the last study drug administration date + REP (16 weeks), or end-of-study date, whichever occurred earlier. Up to a total time frame of 28 weeks (up to week 44).
Description: Double blind period: Safety Analysis Set (SAF): patients who were randomised, and received at least one dose during the trial.
  Open label period: Open label period: Safety analysis set in the open-label treatment period (SAF-OL): This patient set includes all randomized patients who received at least one dose of study drug and received study medication after re-allocation visit (i.e., after Week 16 visit).
Groups:
- Placebo (Week 1-16) and if no Treatment, Week 16-28: Placebo intravenous (i.v.) infusion in the double blind period from baseline to Week 12 (inclusive) - the drug administered 4 times in total. At Week 16 patients were assessed based on their Eczema Area and Severity Index (EASI) score. Patients with EASI>=75 were classified as responders and were followed-up from Week 16 to 28, although receiving no further treatment. Patients with EASI<75 were classified as nonresponders and were offered 600mg Spesolimab treatment in the open label period from Week 16 to 28.
- Spesolimab (Week 1-16) and no Treatment (Week 16-28): 600mg Spesolimab (BI 655130) intravenous (i.v.) infusion in the double blind period from baseline to Week 12 (inclusive) - the drug administered 4 times in total. At Week 16 patients were assessed based on their Eczema Area and Severity Index (EASI) score. Patients with EASI>=75 were classified as responders and were followed-up from Week 16 to 28, although receiving no further treatment. Patients with EASI<75 were classified as non-responders and were offered 600mg Spesolimab treatment in the open label period from Week 16 to 28.
- Spesolimab (Open Label Period, Week 16-44): Following the double blind period (week 0 to 16) patients were assessed based on their Eczema Area and Severity Index (EASI) score, patients with EASI<75 were classified as nonresponders and were offered an open label treatment with 600 mg Spesolimab (BI 655130) i.v. infusion once every 4 weeks from week 16 to 28 (4 treatments in total, last dose at week 28), end of study is at week 44.
Arm/Group | Placebo (Week 1-16) and if no Treatment, Week 16-28 | Spesolimab (Week 1-16) and no Treatment (Week 16-28) | Spesolimab (Open Label Period, Week 16-44)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/33 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/18 | 3/33 | 3/22
Other Adverse Events (participants affected / at risk) | 10/18 | 16/33 | 6/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 1-16) and if no Treatment, Week 16-28 (N=18) | Spesolimab (Week 1-16) and no Treatment (Week 16-28) (N=33) | Spesolimab (Open Label Period, Week 16-44) (N=22)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 1-16) and if no Treatment, Week 16-28 (N=18) | Spesolimab (Week 1-16) and no Treatment (Week 16-28) (N=33) | Spesolimab (Open Label Period, Week 16-44) (N=22)
Eye pruritus (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 2 | 3 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2 | 2
Staphylococcal skin infection (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Blood urine present (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cold urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 7 | 8 | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT03822832/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT03822832/SAP_001.pdf